CLINICAL TRIAL: NCT02049034
Title: The Effect of Lixisenatide on Postprandial Lipid and Glucose Metabolism in Patients with Type 2 Diabetes
Brief Title: Lixisenatide-The Effects on Glucose and Lipid Metabolism in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: LIXISL06684; 2013-002826-22 (EudraCT Number)
Record Dates: First submitted 2013-12-18; First posted 2014-01-29 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1 agonist; Lixisenatide; Postprandial glucose metabolism; Postprandial lipid metabolism; Gastric emptying; Lipoprotein lipase activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide

STUDY DESIGN:
Intervention Model Description: Placebo to IMP (lixisenatide) or IMP (lixisenatide) to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for lixisenatide is supplied as green and purple colored disposable pen-injectors containing 3 mL of a sterile aqueous solution.
  Interventions: Other: Lixisenatide; Other: Placebo
- Lixisenatide (Experimental): Lixisenatide and placebo are considered as investigational medicinal product (IMP). Metformin is not considered an investigational product but concomitant allowed antidiabetic medications.
  Lixisenatide is supplied as disposable pre-filled pen for subcutaneous injection: 10mcg Lixisenatide green pens; 20 mcg Lixisenatide purple pens. Dose titration-10mcg Lixisenatide for 14 days, 20 mcg for 14 days.
  Interventions: Other: Lixisenatide; Other: Placebo

INTERVENTIONS:
Other: Lixisenatide — Lixisenatide and placebo are considered as investigational medicinal product (IMP). Metformin is not considered an investigational product but concomitant allowed antidiabetic medications.
  Lixisenatide is supplied as disposable pre-filled pen for subcutaneous injection: 10mcg Lixisenatide green pens; 20 mcg Lixisenatide purple pens. Dose titration-10mcg Lixisenatide for 14 days, 20 mcg for 14 days.
  Other Names: GLP-1 agonist; Lyxumia
Other: Placebo — Placebo for lixisenatide is supplied as green and purple colored disposable pen-injectors containing 3 mL of a sterile aqueous solution.

SUMMARY:
Glucagon-like-peptide-1 (GLP-1) analogues are a new treatment for type 2 diabetes, which have recently been shown to have beneficial effects on weight, glycaemic control and postprandial triglyceride concentrations. Postprandial hypertriglyceridaemia, which is associated with an increased risk of cardiovascular disease, is a feature of type 2 diabetes. Hypertriglyceridaemia is due to excess triglyceride-rich lipoproteins (TRL) which consist of very low-density lipoproteins, (VLDL) synthesised by the liver which contain the higher molecular weight form of apolipoproteinB (apoB), apoB-100, and chylomicrons which are synthesised in the intestine in response to an intake of dietary fat and contain the lower molecular weight form of apoB, apoB-48. A recent study has shown that GLP-1 receptor signalling is required for the control of postprandial lipoprotein synthesis and secretion in hamsters and mice. GLP-1 was shown to reduce apoB-48 TRL production while a GLP-1 receptor antagonist increased apoB-48 TRL production.

This study will investigate the effect of the GLP-1 analogue lixisenatide compared with placebo, in a double blind crossover study, on postprandial triglyceride metabolism in 12 patients with type 2 diabetes. Chylomicron and VLDL production and clearance rates will be measured in a repeated meal study by labelling apoB-100 and apoB-48 and by labelling triglycerides using stable isotope methodology. Glucose flux in response to a mixed fluid meal will also be investigated using stable isotope methodology. Gastric emptying and post heparin LPL activity will be measured.

The hypothesis is that i] lixisenatide will lower postprandial glycaemia due to a decrease in endogenous glucose output and an increase in glucose clearance by peripheral tissues as a result of an improvement in insulin sensitivity.

DETAILED DESCRIPTION:
GLP-1 analogues are a new treatment for type 2 diabetes, which have recently been shown to have beneficial effects on weight, glycaemic control and postprandial triglyceride concentrations. Postprandial hypertriglyceridaemia, which is associated with an increased risk of cardiovascular disease, is a feature of type 2 diabetes. Hypertriglyceridaemia is due to excess triglyceride-rich lipoproteins (TRL) which consist of very low-density lipoproteins, (VLDL) synthesised by the liver which contain the higher molecular weight form of apolipoproteinB (apoB), apoB-100, and chylomicrons which are synthesised in the intestine in response to an intake of dietary fat and contain the lower molecular weight form of apoB, apoB-48. A recent study has shown that GLP-1 receptor signalling is required for the control of postprandial lipoprotein synthesis and secretion in hamsters and mice. GLP-1 was shown to reduce apoB-48 TRL production while a GLP-1 receptor antagonist increased apoB-48 TRL production.

This study will investigate the effect of the GLP-1 analogue lixisenatide compared with placebo, in a double blind crossover study, on postprandial triglyceride metabolism in 12 patients with type 2 diabetes. Chylomicron and VLDL production and clearance rates will be measured in a repeated meal study (Visits 4 and 8) by labelling apoB-100 and apoB-48 with 1-13C leucine (infusion for 8 hours) and by labelling triglycerides with [1,1,2,3,3-2H5 ]glycerol (as a bolus injection) and 13C triolein. Blood samples will be taken for 4 hours prior to during the 8 hr isotopic infusion to measure the enrichment of apoB-100 and apoB-48 with 1-13C leucine by gas chromatography mass spectrometry.

At Visits 3 and 7, glucose flux in response to a mixed fluid meal containing U-13C glucose will be investigated. Endogenous glucose production will also be measured by infusing [6,6-2H2] glucose for 6hours.

Gastric emptying will be measured by acetaminophen (1000 mg) absorption. Patients will also receive heparin (50U/kg) at the end of the study after 15 minutes a blood sample will be taken to determine post heparin lipoprotein lipase (LPL) activity.

During the study the patients will be asked to monitor their blood glucose for three days with continuous glucose monitoring and to fill in a 7 day food diary.

The hypothesis is that i] lixisenatide will lower postprandial glycaemia due to a decrease in endogenous glucose output and an increase in glucose clearance by peripheral tissues as a result of an improvement in insulin sensitivity.

ii] lixisenatide will reduce postprandial triglycerides due to a decrease in chylomicron production as a result of a direct effect on enterocyte chylomicron assembly and will also reduce VLDL secretion from the liver as a result of an improvement in insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes inadequately controlled by metformin.
* Stable diabetes management over last 3 months: metformin dose unchanged. HbA1c not known to have changed by >0.5% over 3 months.
* Caucasian
* Male
* 40-65 years (inclusive)
* HbA1c 7.5-9.5% (inclusive)
* BMI 27-40 kg/m2 (inclusive)
* Able and willing to self-administer placebo/lixisenatide injection
* Able and willing to perform self-blood glucose monitoring.
* Able and willing to wear a Continuous Glucose Monitoring System (CGMS) for 3 days

Exclusion Criteria:

* Subjects treated with insulin, any oral hypoglycaemic agents (OHA) (other than metformin), any insulin secretagogue or Thiazolidinediones (TZDs)
* A history of heavy alcohol use (>12 to 15 g of alcohol per day)
* Arteriopathy

  * History of significant coronary artery disease (myocardial infarction, surgical or percutaneous [balloon and/or stent] coronary revascularization procedure, or coronary angiography showing at least one stenosis ≥ 50% in a major epicardial artery or branch vessel)
  * Ischemic cerebrovascular disease, including:

    * History of ischemic stroke.
    * History of carotid arterial disease as documented by ≥ 50 % stenosis documented by carotid ultrasound, magnetic resonance imaging or angiography, with or without neurological sequelae.
  * Atherosclerotic peripheral arterial disease, as documented by history of amputation due to vascular disease; history of surgical or percutaneous revascularization procedure; current symptoms of intermittent claudication confirmed by an ankle-brachial pressure index less than 0.9
* Hepatic disease: alanine transaminase (ALT) >3 times upper limit of normal (ULN)
* Renal disease: estimated glomerular filtration rate (Cockroft-Gault equation) less than 40ml/minute.
* Subjects receiving fibrates or weight reducing drugs
* Mental incapacity
* Unwillingness or a language barrier precluding adequate understanding or co-operation
* Fasting plasma triglycerides >4.0 mmol/l
* Systolic blood pressure >160 mmHg on 2 occasions, measured at least 10-minutes apart
* Screening amylase and/or lipase > 3 times ULN or P-calcitonin ≥20 pg/ml (5.9 pmol/L).
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic condition that predisposes to MTC (e.g. multiple endocrine neoplasia syndromes).
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy.
* Any stomach/gastric surgery other than minor endoscopic procedures such as peptic ulcer injection
* Allergic reaction to any GLP-1 receptor agonist or to metacresol.
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting.
* Current smokers
* Subject enrolled in another experimental protocol which involves the use of an investigational drug or device

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose kinetics | Two years
  The study is a double blind cross over study comparing placebo injection with lixisenatide injection. The results will not be known until the investigator is unblinded. An intravenous infusion of [6,6 2H2] glucose will enable the quantification of endogenous hepatic glucose output while addition of [U13C] glucose to a mixed meal will enable the calculation of the contribution of meal derived glucose to postprandial glucose. Enrichment of plasma samples with 2H2 glucose and 13C glucose will be measured by gas chromatography mass spectroscopy (GCMS). Glucose uptake during the postprandial period will then be determined from these measures of glucose output and the glucose concentration at each time point. During this study, gastric emptying will be measured by oral administration of 1000mg acetaminophen.

SECONDARY OUTCOMES:
Postprandial and intestinal triglyceride-rich lipoproteins (TRL) kinetics | Two years
  Triglyceride kinetics in TRLs will be measured by intravenous injection of isotopically labelled glycerol which will be incorporated into nascent triglyceride molecules which is then incorporated into TRL particles (endogenous pathway) and oral administration of 13C triolein which will be incorporated as fatty acids into triglycerides and then become integrated into lipoprotein particles (exogenous pathway). The study uses a feeding protocol which maintains a steady state triglyceride concentration throughout the study. Repeated blood samples will be taken over many hours after administration of the tracers. Hepatic TRL (apoB-100) will be separated from intestinal TRL (ApoB48) using an immunoaffinity method. Measuring the glycerol and 13C oleate enrichments of the triglyceride isolated from lipoproteins, will allow the calculation of the production and clearance rates of triglycerides in both hepatic and intestinal TRLs.

OTHER OUTCOMES:
Post heparin lipoprotein lipase activity | Two years
  A basal sample will be take. Then a heparin will be administered at 50IU/kg. another blood sample will be taken 15 minutes pot heparin injection. Pre and post heparin lipase activity in plasma will be measured using a commercially available kit.
  Both improved β cell function and insulin sensitivity could lead to an increase in LPL activity, increasing the clearance of TRL from the circulation. Improved insulin sensitivity would reduce hepatic TRL synthesis due to direct effects at the liver or indirectly by increasing the insulin sensitivity of lipolysis, thus reducing fatty acid delivery to the liver and intestine. The latter may also impact on intestinal TRL synthesis.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell-Jones, MBBS PhD, Study Chair — Royal Surrey County Hospital NHS Foundation Trust; Margot Umpleby, BA, PhD, Study Director — University of Surrey; Martin Whyte, MBBS, PhD, Principal Investigator — University of Surrey; Fariba Shojaee-Moradie, BSc, PhD, Principal Investigator — Royal Surrey County Hospital & University of Surrey
Locations (1):
- University of Surrey FHMS Diabetes and Metabolic Medicine, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the individual participant data available, however the averaged data has been published .

REFERENCES:
- [Derived] Whyte MB, Shojaee-Moradie F, Sharaf SE, Jackson NC, Fielding B, Hovorka R, Mendis J, Russell-Jones D, Umpleby AM. Lixisenatide Reduces Chylomicron Triacylglycerol by Increased Clearance. J Clin Endocrinol Metab. 2019 Feb 1;104(2):359-368. doi: 10.1210/jc.2018-01176. PMID 30215735
- See also: Whyte MB, Shojaee-Moradie F, Sharaf SE, et al. Lixisenatide Reduces Chylomicron Triacylglycerol by Increased Clearance. J Clin Endocrinol Metab. 2019;104(2):359-368. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6300412/